CLINICAL TRIAL: NCT02843386
Title: Randomized Phase III Study Comparing an Adjuvant Chemotherapy With Fotemustin to Intensive Surveillance in Patients With High Risk Uveal Melanoma
Brief Title: Comparison Between Fotemustin to Intensive Surveillance in Patients With High Risk Uveal Melanoma
Acronym: FOTEADJ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Servier (Industry); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2008-03
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Uveal Melanoma
Keywords: Uveal melanoma; High risk of metastasis; Genomic high risk signature; Adjuvant chemotherapy
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A : Chemotherapy (Experimental): Adjuvant chemotherapy by Fotemustin 100mg/m²
  Interventions: Drug: Adjuvant chemotherapy by Fotemustin
- B : Surveillance (Other): Intensive surveillance
  Interventions: Other: Intensive surveillance

INTERVENTIONS:
Drug: Adjuvant chemotherapy by Fotemustin — Fotemustin is given for 6 cycles :
  * One Induction cycle: Fotemustin 100 mg/m², 1 hour IV infusion, D1D8D15, 5 week rest period, restart on D50.
  * Five Maintenance cycles: Fotemustin 100 mg/m², 1 hour IV infusion, D1-D21.
  Other Names: Fotemustin
  Arms: A : Chemotherapy
Other: Intensive surveillance — Intensive surveillance
  * Total duration: 3 years.
  * liver functional tests/3 months, - liver MRI or CT-scan/6 months, - whole body CT-scan/12 months.
  Other Names: Surveillance
  Arms: B : Surveillance

SUMMARY:
After the local treatment of the primary tumor (protonbeam-therapy, enucleation, external radiotherapy) patients with high risk of metastasis are randomized between:

* Adjuvant chemotherapy with Fotemustin.
* Observation

Both groups are followed during 3 years for Metastasis- Free Survival, safety and tolerance of Fotemustin, quality of life, and Overall Survival.

DETAILED DESCRIPTION:
High risk uveal melanoma is defined by :

* Clinical criteria: Largest Tumor Diameter ≥ 15 mm with extra scleral extension and/or retinal detachment or Largest Tumor Diameter ≥ 18 mm AND/ OR
* Genomic high risk signature (aCGH +/-LOH): Monosomy 3 or partial deletion of 3p associated with any 8 gain.

Treatment schedule :

* Induction: Fotemustin 100 mg/m², D1-D8-D15, 1 hour IV infusion, 1 cycle
* Maintenance : restart on D50, Fotemustine : 100 mg/m², 1 hour IV infusion, D1 D21, 5 cycles.

Both groups are followed during 3 years for Metastasis- Free Survival, safety and tolerance of Fotemustin, quality of life, and Overall Survival.

Note :Based on the second interim analysis showing futility, and no chance to observe any significant statistical difference at the end of the study, the Independent Data Monitoring Committee recommended to stop randomization and amend the protocol to propose an interventional surveillance to high-risk patients as per protocol (April 2016).

ELIGIBILITY:
Inclusion Criteria:

1. High risk uveal melanoma, defined by :

   * Clinical criteria: Largest Tumor Diameter ≥ 15 mm with extrascleral extension and/or retinal detachment or Largest Tumor Diameter ≥ 18 mm AND/OR
   * Genomic high risk signature (cCGH +/- LOH) : Monosomy 3 or partial deletion of 3p and any 8 gain, from enucleation, transscleral or transvitreal samples
2. Age ≥ 18 years and ECOG Performance Status ≤ 2
3. No prior chemotherapy or history of invasive cancer < 5years
4. No metastases
5. Local treatment for the primary tumour (surgery and/or radiotherapy) achieved ≤ 30 days from randomization, chemotherapy to begin within 15 days.

6 - Contraception in women of child-bearing potential

7- Written informed consent

8- Patients with French Social Security in compliance with the French law relating to biomedical research.

Non-Inclusion Criteria:

1. Largest Tumor Diameter < 15 mm or Largest Tumor Diameter 15-18 mm without extrascleral extension and/or retinal detachment, in the absence of genomic alteration as defined per protocol or in the absence of Fine Needle Aspiration biopsy for genomic risk assessment.
2. Contraindication to Fotemustine administration
3. Hematological function : Hb < 10g/dL, absolute neutrophil count < 2,000/mm3, and platelets < 100,000/mm3
4. Biochemistry results :Total bilirubin and AST/ALT > 1,5 UNL (Upper Normal Limit)
5. Creatinine > 1,5 UNL (Upper Normal Limit)
6. Pregnant and/or breastfeeding women.

8 - Previous history of cancer excepting in situ cervical carcinoma or cutaneous basal carcinoma.

7- Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, viral or other hepatitis or cirrhosis, or psychiatric illness/social situation that would interfere with the protocol or limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2009-06-23 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Metastasis-Free survival | 3 years
  Time between patient randomization and metastases occurrence or death

SECONDARY OUTCOMES:
Overall Survival | 3 years
  Time between patient randomization and death
Safety : incidence of Adverse Events and Serious Adverse Events and laboratory abnormalities | 3 years
  using National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) V3
Quality of life assessment | Baseline, 6 months and 3 years
  Using QLQ-C30 questionary.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie PIPERNO-NEUMANN, MD, Principal Investigator — Institut Curie
Locations (6):
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - CHU Nice, Nice
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No